CLINICAL TRIAL: NCT07149259
Title: Assessing the Impact of eSight Go At-Home Usage in Individuals With Visual Impairment
Acronym: eSight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooks Rehabilitation (Other)
Responsible Party: Principal Investigator, Katelyn Jordan, Director of Vision Rehab Services, Brooks Rehabilitation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00085670
Record Dates: First submitted 2025-08-13; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Low Vision Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- At Home Device Utilization (Experimental): eSight Go device will be utilized at home for a total of 4 weeks in environments the participant feels comfortable using it (e.g. home, work, stores).
  Interventions: Device: At Home Use

INTERVENTIONS:
Device: At Home Use — Participants will take the device home for 4 weeks to use in daily living, such as the home and community settings. There will be regular follow-up phone calls once per week from a member of the research team (e.g., an occupational therapist, or low vision therapist) who is familiar with the device to assist with possible troubleshooting as well as device use strategies. The follow up calls will also collect information about device use time and activities. The device will be returned at visit 2.

SUMMARY:
This research aims to test the updated version of Gentex's device, eSight Go, an image enhancing wearable device to assist those with vision impairments limiting activities of daily living.

DETAILED DESCRIPTION:
Subjects will receive introductory training on the controls of the study device at the initial study visit and regular follow-up phone calls once per week from a member of the research staff (e.g., an occupational therapist, or low vision therapist) who is familiar with the study device, to assist with possible troubleshooting as well as device use strategies. You will take the study device home for four weeks to use at school, work, and various daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 90.
* Best-corrected visual acuity between 20/50 to 20/400 in the better eye.
* Subjects who have been diagnosed with an ocular condition causing visual impairment
* Have a functional binocular field of view of at least 20 degrees.
* Visual status stable for at least six months.
* Demonstrate visual benefit from magnification.
* Agree to wear the eSight Go in a variety of situations in the home and community.
* Score ≥ 20 on the Short Orientation-Memory-Concentration Test of Cognitive Impairment (OMCT).
* Subject must be able to provide an informed consent
* Subject must agree to use eSight Eyewear only under conditions that will not jeopardize the safety of either the user or the device.

Exclusion Criteria:

* Participant must not be currently undergoing any medical or surgical procedures resulting in unstable vision.
* Participants who have undergone cataract, refractive, or other surgical procedures related to vision in the six-month period prior to study enrollment.
* Severe (>20/400) visual impairment in the better seeing eye.
* Cognitive limitations (< 20 on OMCT).
* Participants who have undergone any vision-related injections (e.g. anti-VEGF) in the two-month period prior to the study because of active bleeding in the retina. Ongoing anti-VEGF treatments are permitted if the participant is in a "Treat and Extend" or pro re nata ("PRN") disease management, and macula is dry.
* Participants are unable or unwilling to adhere to the examination schedules as they are described in the study protocol. This may also include participants already enrolled, who for whatever reason, have become unable or unwilling to continue the study. This may also include participants for whom the travel time to/from the study site is unacceptable.
* Participants who self-report a history of alcoholism, drug abuse, or psychosis.
* Participants who exhibit clinical evidence of depression, poor motivation, emotional or intellectual problems, or any other conditions which would likely limit validity of consent or appropriate responses to participate in the study or who are deemed unsuitable psychologically or physiologically for study participation by the investigator.
* Participants who may have a conflict of interest with eSight Corp, which could reasonably influence their participation in the study.
* Refractive error outside the range correctable by lens inserts in the device (> +/-8.00 D sph or -4.00 cyl)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Acuity | Pre-intervention and post-intervention at 4 weeks
  Early Treatment Diabetic Retinopathy Study Chart (ETDRS) assessing visual acuity. A lower logMAR value indicates an improved score.
Change in Reading Performance | Pre-intervention and post-intervention at 4 weeks
  Minnesota Low Vision Reading Test assessing reading performance. A lower logMAR value indicates an improved score.

SECONDARY OUTCOMES:
Change in Mobility | Pre-intervention and post-intervention at 4 weeks
  Dynamic Gait Index (DGI) assessing the ability of the participant to maintain walking balance. 8 items are scored on a scale of 0 to 4, where 0=severe impairment, 1=moderate impairment, 2=mild impairment, and 3=normal. An increase in score reflects an improvement in mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn Jordan, D.O., Principal Investigator — Brooks Rehabilitation
Locations (1):
- Brooks Rehabilitation, Jacksonville, Florida, United States

DOCUMENTS (1):
  • Study Protocol (2025-04-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT07149259/Prot_000.pdf